CLINICAL TRIAL: NCT03595358
Title: A Prospective Multi-Centre Study of the Ellume·Lab Flu A+B Test and the Ellume Home Flu Test Performance Versus Viral Culture and Reverse Transcriptase Polymerase Chain Reaction
Brief Title: Ellume·Lab Flu A+B Test and the Ellume Home Flu Test Performance Versus Viral Culture and Reverse Transcriptase Polymerase Chain Reaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ellume Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IE-FLU-AUS-1801
Record Dates: First submitted 2018-07-11; First posted 2018-07-23 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm (Experimental): Ellume Home Flu Test and ellume.lab Flu A+B Test
  Upper respiratory tract samples from participants will be tested with:
  Ellume Home Flu Test; ellume.lab Flu A+B Test; Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) and viral culture.
  Interventions: Diagnostic Test: Ellume Home Flu Test; Diagnostic Test: ellume.lab Flu A+B Test; Diagnostic Test: Reverse Transcriptase Polymerase Chain Reaction (RT-PCR); Diagnostic Test: Viral culture

INTERVENTIONS:
Diagnostic Test: Ellume Home Flu Test — The Ellume Home Flu Test is a rapid in vitro diagnostic test for the detection of influenza A or influenza B in nasal swab samples.
Diagnostic Test: ellume.lab Flu A+B Test — The ellume.lab Flu A+B Test is a rapid in vitro diagnostic test intended to be used at point-of-care for the detection of influenza A or influenza B in nasal swab samples.
Diagnostic Test: Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) — Reverse Transcriptase Polymerase Chain Reaction (RT_PCR) is a molecular diagnostic technique for the detection and identification of influenza viruses, both for clinical samples and isolates. The Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) allows template viral RNA to be reverse transcribed producing complementary DNA (cDNA) which can then be amplified and detected.
Diagnostic Test: Viral culture — Nasopharyngeal samples will be inoculated into appropriate culture media for influenza viral culture. In this test, the virus is actually grown and further identified in the laboratory as influenza A or B.

SUMMARY:
The primary purpose of the study is to validate the sensitivity and specificity of the Ellume Home Flu Test and the ellume.lab Flu A+B Test in detecting influenza A and influenza B as compared to reverse transcriptase polymerase chain reaction (RT-PCR)

Secondary aims are to:

Validate the sensitivity and specificity of the Ellume Home Flu Test and the ellume.lab Flu A+B Test in detecting influenza A and influenza B as compared to viral culture; Evaluate the participant's satisfaction with the convenience and ease of use of the Ellume Home Flu Test; Evaluate the participant's interpretation of the Ellume Home Flu Test results compared to the interpretation by site staff; Evaluate the operator's satisfaction and ease of use of the ellume·lab Flu A+B Test.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged ≥ 2 years; and
* Fever ≥ 37.8° C (100° F) at presentation or history or parent/guardian-reported history of fever ≥ 37.8° C or feeling feverish within 24 hours of presentation; and
* Rhinorrhea; and
* ≤ 72 hours from onset of ILI symptoms; and
* Participant (or parent/legal guardian) capable and willing to give informed consent/assent; and
* Participant (or parent/legal guardian) able to read and write in English.

Exclusion Criteria:

* Participants aged < 2 years.
* Participants who have undergone treatment with Tamiflu (oseltamivir), Relenza (zanamivir) or Symmetral (amantadine) within the previous 7 days;
* Participants who have been vaccinated by means of an Influenza nasal spray/mist vaccine within the previous 7 days;
* Participants who have had a nose bleed within the past 30 days;
* Participants who have had recent craniofacial injury or surgery, including surgery to correct deviation of the nasal septum, within the previous 6 months;
* Participants currently enrolled in another clinical trial or used any investigational device within 30 days preceding informed consent.
* Participants previously enrolled in IE-FLU-AUS-1801;
* Participants 18 years of age or older unable to understand English and consent to participation;
* Parent/legal guardian of participants < 18 years of age unable to understand English and consent to participation of child.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2018-11-16 (Actual)

PRIMARY OUTCOMES:
Of participants positive for influenza A by Reverse Transcriptase Polymerase Chain Reaction (RT-PCR), the percentage who are positive for influenza A by Ellume Home Flu Test. | 1 day
  Establish sensitivity against a gold standard. Report as a percentage of participants with 96% confidence intervals.
Of participants positive for influenza A by Reverse Transcriptase Polymerase Chain Reaction (RT-PCR), the percentage who are positive for influenza A by ellume.lab Flu A+B Test. | 1 day
  Establish sensitivity against a gold standard. Report as a percentage of participants with 96% confidence intervals.
Of participants negative for influenza A by Reverse Transcriptase Polymerase Chain Reaction (RT-PCR), the percentage who are negative for influenza A by Ellume Home Flu Test. | 1 day
  Establish specificity against a gold standard. Report as a percentage of participants with 96% confidence intervals.
Of participants negative for influenza A by Reverse Transcriptase Polymerase Chain Reaction (RT-PCR), the percentage who are negative for influenza A by ellume.lab Flu A+B Test. | 1 day
  Establish specificity against a gold standard. Report as a percentage of participants with 96% confidence intervals.
Of participants positive for influenza B by Reverse Transcriptase Polymerase Chain Reaction (RT-PCR), the percentage who are positive for influenza B by Ellume Home Flu Test. | 1 day
  Establish sensitivity against a gold standard. Report as a percentage of participants with 96% confidence intervals.
Of participants positive for influenza B by Reverse Transcriptase Polymerase Chain Reaction (RT-PCR), the percentage who are positive for influenza B by ellume.lab Flu A+B Test. | 1 day
  Establish sensitivity against a gold standard. Report as a percentage of participants with 96% confidence intervals.
Of participants negative for influenza B by Reverse Transcriptase Polymerase Chain Reaction (RT-PCR), the percentage who are negative for influenza B by Ellume Home Flu Test. | 1 day
  Establish specificity against a gold standard. Report as a percentage of participants with 96% confidence intervals.
Of participants negative for influenza B by Reverse Transcriptase Polymerase Chain Reaction (RT-PCR), the percentage who are negative for influenza B by ellume.lab Flu A+B Test. | 1 day
  Establish specificity against a gold standard. Report as a percentage of participants with 96% confidence intervals.

SECONDARY OUTCOMES:
Of participants positive for influenza A by viral culture, the percentage who are positive for influenza A by Ellume Home Flu Test. | 1 day
  Establish sensitivity against a gold standard. Report as a percentage of participants with 96% confidence intervals.
Of participants positive for influenza A by viral culture, the percentage who are positive for influenza A by ellume.lab Flu A+B Test. | 1day
  Establish sensitivity against a gold standard. Report as a percentage of participants with 96% confidence intervals.
Of participants negative for influenza A by viral culture, the percentage who are negative for influenza A by Ellume Home Flu Test. | 1 day
  Establish specificity against a gold standard. Report as a percentage of participants with 96% confidence intervals.
Of participants negative for influenza A by viral culture, the percentage who are negative for influenza A by ellume.lab Flu A+B Test. | 1 day
  Establish specificity against a gold standard. Report as a percentage of participants with 96% confidence intervals.
Of participants positive for influenza B by viral culture, the percentage who are positive for influenza B by Ellume Home Flu Test. | 1 day
  Establish sensitivity against a gold standard. Report as a percentage of participants with 96% confidence limits.
Of participants positive for influenza B by viral culture, the percentage who are positive for influenza B by ellume.lab Flu A+B Test. | 1 day
  Establish sensitivity against a gold standard. Report as a percentage of participants with 96% confidence intervals.
Of participants negative for influenza B by viral culture, the percentage who are negative for influenza B by Ellume Home Flu Test. | 1 day
  Establish specificity against a gold standard. Report as a percentage of participants with 96% confidence intervals.
Of participants negative for influenza B by viral culture, the percentage who are negative for influenza B by ellume.lab Flu A+B Test. | 1 day
  Establish specificity against a gold standard. Report as a percentage of participants with 96% confidence intervals.
Percent of participants who correctly interpret the result of the Ellume Home Flu Test | 1 day
  Agreement between trained staff and participants. Report as a percentage of participants with 96% confidence limits.
Scores from questionnaire to assess ease of use, comfort and convenience of the Ellume Home Flu Test. | 1 day
  The ease of use questionnaire will provide total number of responses to each question and the percentage of participants selecting each response (on a 5 point Likert scale).
Scores from questionnaire to assess ease of use and convenience of the ellume.lab Flu A+B Test. | 1 day
  The ease of use questionnaire will provide total number of responses to each question and the percentage of participants selecting each response (on a 5 point Likert scale).

CONTACTS AND LOCATIONS:
Locations (1):
- Paratus Clinical Kanwal Trial Clinic, Kanwal, New South Wales, Australia